CLINICAL TRIAL: NCT06856356
Title: Comparison of Clinical Efficacy and Safety of Robot-assisted Total Knee Arthroplasty and Conventional Total Knee Arthroplasty: a Randomized Controlled Study
Brief Title: Clinical Efficacy and Safety of Robot-assisted Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJS2023-1-18(WK)
Record Dates: First submitted 2024-08-14; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis, Knee
Keywords: total knee arthroplasty; robot-assisted; alignment; satisfication; complication
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors are independent of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robot-assisted total knee arthroplasty (Experimental): Using an orthopedic joint surgery navigation system to assist total knee replacement
  Interventions: Procedure: Robot-assisted surgery
- Conventional total knee arthroplasty (Active Comparator): Using a conventional 4-in-1 osteotomy guide for total knee replacement
  Interventions: Procedure: Conventional total knee arthroplasty

INTERVENTIONS:
Procedure: Robot-assisted surgery — Orthopedic surgeons perform total knee arthroplasty using an orthopedic joint surgery navigation system
  Arms: Robot-assisted total knee arthroplasty
Procedure: Conventional total knee arthroplasty — Orthopedic surgeons perform total knee arthroplasty using a 4 in 1 osteotomy guide
  Arms: Conventional total knee arthroplasty

SUMMARY:
The purpose of this clinical trial is to understand the application value of the Orthopedic Joint Surgery Navigation System in assisting surgeons to accurately place prosthetic components in adult knee replacement surgery. It will also confirm its effectiveness and safety in clinical application.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to understand the application value of the Orthopedic Joint Surgery Navigation System in assisting surgeons to accurately place prosthetic components in adult knee replacement surgery. It will also confirm its effectiveness and safety in clinical application. The main questions it aims to answer are:

Does the Orthopedic Joint Surgery Navigation System improve the accuracy of prosthetic component placement in knee replacement surgery? Is the Orthopedic Joint Surgery Navigation System superior to traditional total knee replacement What medical problems do participants encounter when taking medication ABC? Researchers will compare the Orthopedic Joint Surgery Navigation System with traditional total knee replacement surgery (using a "four-in-one" osteotomy guide) to see if the Orthopedic Joint Surgery Navigation System is superior to traditional total knee replacement in terms of prosthesis three-dimensional position, force alignment, patient satisfaction, functional scores, complications, etc.

Participants will:

End-stage knee osteoarthritis patients receive total knee replacement with the Orthopedic Joint Surgery Navigation System or traditional total knee replacement surgery Visit the clinic for examination and testing every 3 months Record their imaging data, satisfaction, functional scores, complications, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in the trial and sign the informed consent form;
2. Aged 18 to 80 years old (inclusive), regardless of gender;
3. Patients who need total knee replacement surgery;
4. Those who can communicate well with the researchers and comply with the trial requirements.

Exclusion Criteria:

1. Patients who are allergic to the drugs used in this trial or the implant materials;
2. Patients with immature bone development;
3. Patients with active infection;
4. Patients with neuropathy of the knee joint;
5. Patients with poor bone quality that is not conducive to prosthesis fixation;
6. Patients with general conditions or concomitant diseases that make it difficult for people to tolerate surgery;
7. Patients with insufficient quadriceps muscle strength;
8. Patients with insufficient skin coverage near the surgical site and intolerance to surgery;
9. Patients with severe femoral or tibial deformities and other severe deformities outside the joint;
10. Patients with metal implants in the joint surgical area that affect the execution of the surgical plan;
11. Pregnant or lactating women;
12. Patients with severe epilepsy or mental illness;
13. Patients with alcohol dependence or drug addiction;
14. Patients with severe coagulation disorders;
15. Patients who have participated in or are participating in other clinical trials within one month of enrollment;
16. Patients who are considered by the researchers to be unsuitable for participating in this clinical trial for other reasons. Those who meet any of the above exclusion criteria need to be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative patient satisfaction | Month 1, Month 3, Month 6, Month 12, Month 24
  Use a questionnaire to investigate patients' satisfaction with their knee joint after surgery
Forgotten Joint Scores | Month 1, Month 3, Month 6, Month 12, Month 24
  The Forgotten Joint Score (FJS) is a validated patient-reported outcome measure (PROM) tool designed to assess artificial prosthesis awareness during daily activities following total knee arthroplasty.The total score is 100 points. The higher the score, the better the degree of forgetfulness of the artificial joint.
WOMAC score | Month 1, Month 3, Month 6, Month 12, Month 24
  Use WOMAC scoring scale to assess the condition of the knee joint. The WOMAC score consists of 24 items with a total score of 100. The higher the score, the more severe the limitation of joint function.
Knee Society Score | Month 1, Month 3, Month 6, Month 12, Month 24
  The KSS score was assessed using the American Knee Society scoring criteria.The full score is 100 points. The higher the score, the better the patient's knee function.

SECONDARY OUTCOMES:
SF-12 | Month 1, Month 3, Month 6, Month 12, Month 24
  The health status of patients was assessed using the SF-12 health-related quality of life scale. The higher the score, the better the quality of life.
visual analogue scale score | Month 1, Month 3, Month 6, Month 12, Month 24
  Visual analogue scale (VAS) for pain assessment。0 means no pain, 10 means the most painful, the higher the value, the higher the pain level of the patient
Range of motion | Month 1, Month 3, Month 6, Month 12, Month 24
  Physical examination to assess the knee's range of motion
Hip-knee-ankle angle | postoperative Day 1-3
  Measuring Hip-knee-ankle angle in radiology
Complication | Month 1, Month 3, Month 6, Month 12, Month 24
  Record the patient's postoperative complications. For example, Persistent pain, fracture, superficial local infection, infection, thromboembolism.

OTHER OUTCOMES:
mLDFA | preoperative Day 1-3, postoperative Day 1-3
  the lateral angle between the mechanical axis of the femur and the tangent of the distal end of the femoral prosthesis. The target value is 90°. >90° is varus, and <90° is valgus. Varus or valgus exceeding 3° is defined as femoral prosthesis position deviation.
mMPTA | preoperative Day 1-3, postoperative Day 1-3
  medial angle between the mechanical axis of the tibia and the tangent of the tibial prosthesis, the target value is 90°, <90° is varus, >90° is valgus, and valgus exceeding 3° is defined as tibial prosthesis position deviation
Femoral prosthesis flexion angle (α angle) | preoperative Day 1-3, postoperative Day 1-3
  on the standard lateral knee X-ray, the angle between the anatomical axis of the distal femur and the vertical line of the distal femoral prosthesis
Tibial posterior tilt angle (β angle): | preoperative Day 1-3, postoperative Day 1-3
  on the standard lateral knee X-ray, the angle between the anatomical axis of the tibia and the lower surface of the tibial prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Zhu, M.D, Principal Investigator — The First Affiliated Hospital of USTC
Locations (1):
- the first affiliated hospital of USTC, Hefei, Anhui, China